CLINICAL TRIAL: NCT05133635
Title: Comparison of the Treatment Efficacy of High-Dose Corticosteroid and Tocilizumab During Clinical Worsening in Patients With COVID-19 Pneumonia
Brief Title: High-Dose Corticosteroid or Tocilizumab for Clinical Worsening of COVID-19
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: A recent study suggested a new corticosteroid regime for intensive care unit patients.
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Ruslan Abdullayev, Assist. Prof., Marmara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Steroid/Toci COVID-19
Record Dates: First submitted 2021-01-11; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: COVID-19 Virus Infection; Cytokine Storm; Corticosteroid; Tocilizumab
MeSH Terms: conditions — COVID-19; Cytokine Release Syndrome | interventions — Methylprednisolone; Adrenal Cortex Hormones; tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pulse methylprednisolone (Active Comparator): 250 mg methylprednisolone for 3 days
  Interventions: Drug: Methylprednisolone
- Tocilizumab (Active Comparator): Tocilizumab 400-800 mg for one time
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Methylprednisolone — Patients with the clinical and laboratory diagnosis of cytokine storm will receive methylprednisolone 250 mg for 3 days.
  Other Names: Corticosteroid
  Arms: Pulse methylprednisolone
Drug: Tocilizumab — Patients with the clinical and laboratory diagnosis of cytokine storm will receive tocilizumab 400-800 mg for one time.
  Arms: Tocilizumab

SUMMARY:
COVID-19 pandemic has spread all over the world, and hospitalization of the patients with COVİD-19 Pneumonia has become a great burden to the Intensive Care Units. Unfortunately there is still no curative method for the disease yet. Intensive Care Units provide general care for the patients; including oxygen therapy, maintenance of the organ systems (e.g., cardiovascular, renal), nutrition, antibiotic therapy for secondary infections, and etc.

One of the major problems in COVID-19 is macrophage activation syndrome, also known as cytokine storm. It stems from exaggerated inflammatory response, which causes increased cytokine release and results in clinical deterioration of the patients. Many drugs have been used to prevent this exaggerated inflammation, like corticosteroids, interleukin (IL) receptor blockers, plasma exchange, etc.

In this study our aim is to investigate the effectiveness of high dose corticosteroid (methylprednisolone 250 mg for 3 days) and an IL-6 receptor antagonist (tocilizumab) in the treatment of the cytokine storm of the COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with COVID-19 Pneumonia treated in the Intensive Care Unit
* Clinical deterioration during intensive care follow-up
* First 14 days from the COVID-19 diagnosis

Exclusion Criteria:

* More than 14 days passed from the COVID-19 diagnosis
* Clinical and laboratory signs of secondary bacterial infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Clinical condition | Next 7 days of the intervention.
  Arterial oxygen partial pressure of the patient will be observed.
Blood analysis | Next 7 days of the intervention.
  Acute phase reactants (C-reactive protein, procalcitonin, ferritin, fibrinogen), will be investigated.

SECONDARY OUTCOMES:
Hospital stay | Until the hospital discharge.
  Hospital stay period of the patients will be observed.
Mortality | Not relevant
  Mortality of the patients will be observed.

CONTACTS AND LOCATIONS:
Overall Officials: Ruslan Abdullayev, Principal Investigator — Marmara University

IPD SHARING:
Plan to Share IPD: No